CLINICAL TRIAL: NCT00766103
Title: The Effects of PaCO2 Levels on Cerebral Metabolism and Perfusion During Induced Hypothermia.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tampere University Hospital (Other)
Responsible Party: Principal Investigator, Patrik Falkenbach, Md, Tampere University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: R06213
Record Dates: First submitted 2008-10-02; First posted 2008-10-03 (Estimated); Last update posted 2016-10-21 (Estimated); Status verified 2016-10

CONDITIONS: Cerebral Metabolism and Perfusion
Keywords: Cerebral metabolism, perfusion, induced hypothermia

ARMS (1):
- crossover: hypo- and hypercarbia (Other)
  Interventions: Other: mild hypo- and hyperventilation

INTERVENTIONS:
Other: mild hypo- and hyperventilation — induction of mild hypo- and hypercarbia

SUMMARY:
Incidence of hypo- and hypercarbia during induced hypothermia after cardiac arrest is high. The original report from HACA-group reported that hypothermia treated patients had improved survival and neurological outcome. Suprisingly, in that trial normocarbia was not achieved even though the aim was set for ventilatory support as normoventilation. This study aims to investigate the effects of mild hypo- and hypercarbia on cerebral perfusion (blood flow, intracranial pressure) and metabolism (microdialysate metabolites). We hypothesize that uncontrolled ventilatory suppport may render the patients in risk of exacerbation of neuronal damage, conversely, further improvement in outcome may be achieved with succesfull ventilatory management. We intend to enroll 10 out-of-hospital cardiac arrest patients succesfully resuscitated and subsequently treated with controlled hypothermia for 24 hours. The patients in need of anticoagulation are excluded. We plan to induce mild hypocarbia and hypercarbia during and after induced hypothermia. Metabolic and perfusion data are collected with clinically used methods such as transcranial doppler, intracranial pressure measurement, near infrared spectroscopy, jugular bulb, intracerebral microdialysis).

ELIGIBILITY:
Inclusion Criteria:

succesfull resuscitation of out of hospital cardiac arrest, primary rhytm shockable

Exclusion Criteria:

* known coagulopathy, need of anticoagulation therapy, need of interventional cardiological procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2006-12; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
surrogate physiological endpoints | 60minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Critical Care Medicine Research Group/ department of intensive care, Tampere, Pirkanmaa, Finland

REFERENCES:
- See also: Tampere University Hospital (Pirkanmaa hospital district) home page (in English) — http://www.pshp.fi/default.aspx?contentlan=2
- See also: Home page of the Science Center of Tampere University Hospital (in Finnish) — http://www.pshp.fi/default.aspx?nodeid=10066&contentlan=1